CLINICAL TRIAL: NCT06986135
Title: The Effect of Breathing Interventions on Biomarkers of Stress and Cognitive Performance Following a Psychologically Stressful Task
Brief Title: The Effect of Breathing on Cognitive Performance and Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas State University (Other)
Collaborators: Texas State University, San Marcos (Other)
Responsible Party: Principal Investigator, Matt McAllister, Associate Professor, Texas State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: IRB #9665
Record Dates: First submitted 2025-05-07; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Stress; Acute Stress Reaction; Breathing Techniques; Cognitive Performance
Keywords: Stress; Trier Social Stress Test; Acute Stress; Breathing Technique; Box Breathing; Cognitive Performance; Biomarkers
MeSH Terms: conditions — Stress Disorders, Traumatic, Acute

STUDY DESIGN:
Intervention Model Description: Subjects were randomly assigned to one of three groups, between and within subject analysis occurred.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Box Breathing group (Experimental): Group to be assigned box breathing.
  Interventions: Other: Box Breathing
- Prolonged Exhalation Breathing assignment group (Experimental): Breathing group to be assigned the prolonged exhalation intervention.
  Interventions: Other: Prolonged Exhalation
- Placebo (normal breathing) group (Placebo Comparator): This group is not assigned a breathing technique, and acts as a placebo.
  Interventions: Other: Normal Breathing

INTERVENTIONS:
Other: Box Breathing — Box breathing consisted of a 4 second inhale, 4 second hold, 4 second exhale, 4 second hold; for 4 minutes.
  Arms: Box Breathing group
Other: Prolonged Exhalation — Prolonged Exhalation consisted of a deep, 3 second inhale, followed by a slow 6 second exhale through pursed lips, once every 30 seconds for 4 minutes.
  Arms: Prolonged Exhalation Breathing assignment group
Other: Normal Breathing — This was the placebo, normal breathing group was instructed to breath as they normally would for the entirety of the 4 minute period.
  Arms: Placebo (normal breathing) group

SUMMARY:
The purpose of this study is to determine the effectiveness of different breathing techniques on biomarkers of stress and cognitive performance following the Trier Social Stress Test.

DETAILED DESCRIPTION:
This study examined the effect of three various breathing techniques (i.e., normal breathing, prolonged exhalation, and box breathing) on biomarkers of stress and mental performance after the Trier Social Stress Test (TSST). The TSST has been shown to result in significant increases in psychological and physiological stress markers. Therefore, the goal of this study was to examine potential interventions to mitigate the effects of this psychological stressor while maintaining increased cognitive performance. Moreover, previous literature has shown various effects of breathing interventions, therefore, the investigators wished to further validate breathing techniques as an effective tool to mitigate stress and increase cognitive performance. The data from this research provided insight to real life events, allowing for a principal understanding of how to reduce stress, focused at first responder populations.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy
* Between the ages of 18-39,
* Student at Texas State.

Exclusion Criteria:

* Any known cardiovascular or metabolic disease
* Consuming any medication for psychiatric disorders (i.e., anxiety, depression, ADHD)
* Being diagnosed with any psychiatric or physical conditions
* Any major stressors in the last 30 days (i.e., birth of a child, abortion, divorce).

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Cognitive Challenge | 20 minutes prior to TSST start and immediately post TSST.
  Subjects participated in a 1 minute familiarization for the Stroop Color Word Challenge, followed by a full 2 minute Stroop Color Word challenge. Immediately following the Stroop, subjects then participated in a 2 minute mental arithmetic. The Stroop consisted of conflicting color-word fonts, and the subject had to choose the correct font color: subjects had .5 seconds to respond to each answer utilizing a color coordinated keypad. The mental arithmetic consisted of a series of mathematical problems (i.e., one, two, or three digit addition and subtraction). If subjects got an answer wrong for the mental math, a buzzer would sound.
Heart Rate | HR was recorded 4 times, during each saliva sample collection period
  Heart rate was recorded immediately prior to each saliva sample using the same tools to record the HRV measure. The Polar H10 and HRVTrace app was utilized to record a Heart rate measure 4 times throughout the study.
State Anxiety Inventory (SAI) | Timepoint 1-4, 40 minutes pre, 10 minutes pre, immediately post, 25 minutes post.
  The SAI is a 6 question survey on a 24 point scale, asking the subject to record how they feel. Questions asked were "I am calm", "I am tense", "I am worried", "I am relaxed", etc. Subjects were asked to fill this out 4 times throughout the study, alongside the HR and saliva samples.
Heart rate variability | HRV was recorded immediately following the 2nd, 3rd, and 4th saliva samples.
  Heart Rate Variability (HRV) was measured three times over the course of the study in order to measure responses to stress. A Polar H10 monitor was used, alongside the HRVTrace app to record the three measures. Each HRV measurement was 7 minutes, and required the subjects to sit quietly and watch a standardized nature video.
Secretory Immunoglobin-A | 40 minutes prior to modified TSST start, 10 minutes prior to modified TSST start, immediately post modified TSST, and 25 minutes post TSST
  SIgA is a marker of immune function and salivary SIgA concentrations tend to increase when exposed to stress
Salivary Alpha Amylase | 40 minutes prior to modified TSST start, 10 minutes prior to modified TSST start, immediately post modified TSST, and 25 minutes post TSST
  salivary alpha amylase is an enzyme involved in digestive processes. Amylase concentration in saliva have been shown to reflect sympathetic stress. Thus, as sympathetic stress increases, salivary amylase concentrations tend to increase.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas State University, Metabolic & Applied Physiology Lab, San Marcos, Texas, United States

IPD SHARING:
Plan to Share IPD: No
IRB at Texas State does not allow the sharing of individual data, and all data has already been made unidentifiable for this study.

REFERENCES:
- [Background] Kotlyar M, Donahue C, Thuras P, Kushner MG, O'Gorman N, Smith EA, Adson DE. Physiological response to a speech stressor presented in a virtual reality environment. Psychophysiology. 2008 Nov;45(6):1034-7. doi: 10.1111/j.1469-8986.2008.00690.x. Epub 2008 Sep 4. PMID 18778321
- [Background] Allen AP, Kennedy PJ, Dockray S, Cryan JF, Dinan TG, Clarke G. The Trier Social Stress Test: Principles and practice. Neurobiol Stress. 2016 Nov 12;6:113-126. doi: 10.1016/j.ynstr.2016.11.001. eCollection 2017 Feb. PMID 28229114
- [Background] Matsumoto T, Masuda T, Hotta K, Shimizu R, Ishii A, Kutsuna T, Yamamoto K, Hara M, Takahira N, Matsunaga A. Effects of prolonged expiration breathing on cardiopulmonary responses during incremental exercise. Respir Physiol Neurobiol. 2011 Sep 15;178(2):275-82. doi: 10.1016/j.resp.2011.06.025. Epub 2011 Jul 7. PMID 21763472
- [Background] Narkiewicz K, van de Borne P, Montano N, Hering D, Kara T, Somers VK. Sympathetic neural outflow and chemoreflex sensitivity are related to spontaneous breathing rate in normal men. Hypertension. 2006 Jan;47(1):51-5. doi: 10.1161/01.HYP.0000197613.47649.02. Epub 2005 Dec 12. PMID 16344363
- [Background] Ntovas P, Loumprinis N, Maniatakos P, Margaritidi L, Rahiotis C. The Effects of Physical Exercise on Saliva Composition: A Comprehensive Review. Dent J (Basel). 2022 Jan 5;10(1):7. doi: 10.3390/dj10010007. PMID 35049605
- [Background] Dillard CC, Martaindale H, Hunter SD, McAllister MJ. Slow Breathing Reduces Biomarkers of Stress in Response to a Virtual Reality Active Shooter Training Drill. Healthcare (Basel). 2023 Aug 21;11(16):2351. doi: 10.3390/healthcare11162351. PMID 37628548
- [Background] Kim HG, Cheon EJ, Bai DS, Lee YH, Koo BH. Stress and Heart Rate Variability: A Meta-Analysis and Review of the Literature. Psychiatry Investig. 2018 Mar;15(3):235-245. doi: 10.30773/pi.2017.08.17. Epub 2018 Feb 28. PMID 29486547